CLINICAL TRIAL: NCT02485041
Title: An Open Label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetic Interaction of Dapoxetine 30 mg and Mirodenafil 100 mg in Healthy Male Volunteers
Brief Title: Pharmacokinetic Interaction Study of Dapoxetine 30mg and Mirodenafil 100mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SID123_DDI_I_2014
Record Dates: First submitted 2015-06-12; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Drug Interaction Potentiation
Keywords: Dapoxetine; Mirodenafil; DDI study
MeSH Terms: interventions — dapoxetine; mirodenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- M→D→D+M (Experimental): Mirodenafil(M) in period 1, Dapoxetine(D) in period 2, Dapoxetine+Mirodenafil(D+M) in period 3
  Interventions: Drug: Dapoxetine 30mg; Drug: Mirodenafil 100mg
- M→D+M→D (Experimental): Mirodenafil(M) in period 1, Dapoxetine+Mirodenafil(D+M) in period 2, Dapoxetine(D) in period 3
  Interventions: Drug: Dapoxetine 30mg; Drug: Mirodenafil 100mg
- D→M→D+M (Experimental): Dapoxetine(D) in period 1, Mirodenafil(M) in period 2, Dapoxetine+Mirodenafil(D+M) in period 3
  Interventions: Drug: Dapoxetine 30mg; Drug: Mirodenafil 100mg
- D→D+M→M (Experimental): Dapoxetine(D) in period 1, Dapoxetine+Mirodenafil(D+M) in period 2, Mirodenafil(M) in period 3
  Interventions: Drug: Dapoxetine 30mg; Drug: Mirodenafil 100mg
- D+M→M→D (Experimental): Dapoxetine+Mirodenafil(D+M) in period 1, Mirodenafil(M) in period 2, Dapoxetine(D) in period 3
  Interventions: Drug: Dapoxetine 30mg; Drug: Mirodenafil 100mg
- D+M→D→M (Experimental): Dapoxetine+Mirodenafil(D+M) in period 1, Dapoxetine(D) in period 2, Mirodenafil(M) in period 3
  Interventions: Drug: Dapoxetine 30mg; Drug: Mirodenafil 100mg

INTERVENTIONS:
Drug: Dapoxetine 30mg — Tablet, Orally administered
Drug: Mirodenafil 100mg — Table, Orally administered

SUMMARY:
Healthy male volunteers were administered alone and in combination with dapoxetine 30mg mirodenafil 100mg for three times, respectively and the pharmacokinetic interaction was compared between the two drugs.

DETAILED DESCRIPTION:
Healthy male volunteers were randomized into one group among 6 sequential groups and were administered alone or in combination with dapoxetine 30mg mirodenafil 100mg in each period. Bloods were obtained at each time for pharmacokinetic analysis. Safety evaluation was also done during entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged between 19 and 55
* Body mass index (BMI) in the range of 19 to 27 kg/m2
* Understand the requirements of the study and voluntarily consent to participate in the study
* Available for the entire study period

Exclusion Criteria:

* Subject has a history such as liver diseases, kidneys, digestive system, respiratory system, endocrine system, nervous psychiatric, blood, cancer, cardiovascular diseases
* Subject with clinically significant vital signs (sitting position blood pressure) (90 mmHg > systolic blood pressure ≥ 140 mmHg, 60 mmHg > diastolic blood pressure ≥ 90 mmHg)
* History of drug abuse
* History of caffeine, alcohol, smoking abuse

  * caffeine(coffee,tea,coke)> 4cups/day
  * smoking > 10 cigarettes/day
  * alcohol > 140g/week
* Consumption of any grapefruit or grapefruit-containing juices over 1 cup a day
* Previously donate whole blood within 60 days or component blood within 30 days
* Subject has taken drugs which affects the ADME of investigational products
* Subject with known for hypersensitivity reactions to mirodenafil/ dapoxetine or other drugs
* Inadequate laboratory test result:

  * AST(SGOT) or ALT(SGPT) or total bilirubin > 1.5 x upper limit of normal range
* Subject considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cmax | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Cmax of dapoxetine and mirodenafil
Area Under Curve (AUC) | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  AUC of dapoxetine and mirodenafil

SECONDARY OUTCOMES:
Tmax | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
t1/2 | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
CL/F | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
Vd/F | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
Number of Participants with Adverse events | During 22 days from first administration of period 1
  Incidence rate of Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, PhD, Principal Investigator — Chonbuk National University Hospital